CLINICAL TRIAL: NCT03639272
Title: Long-term Radiographic and Clinical-functional Outcomes of Isolated, Displaced, Closed Talar Neck and Body Fractures Treated by Open Reduction Iternal Fixation: the Timing of Surgical Management.
Brief Title: Treatment of Talus Fractures: a Retrospective Study
Acronym: TTF2017
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Carlo Biz, Orthopedic surgeon, Assistant Professor, University of Padova
Other Study IDs: 4065/AO/17
Record Dates: First submitted 2018-07-31; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Talus Fracture
Keywords: talar fractures; talar neck fractures;; talar body fractures;; talus;; ORIF;; screw fixation.
MeSH Terms: interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: open reduction and internal fixation (ORIF). — Depending on the fracture location, a single anteromedial or anterolateral approach was carried out. The fracture site was cleaned to make it visible, allowing anatomical reduction. Subsequently, fixation of provisional fragments was achieved using temporary Kirschner wires under radiographic guidance. Having obtained satisfactory reduction as seen with the radiographic intensifier, definitive fixation of the main bone fragments was carried out using two or more 3.5 mm titanium cannulated screws or 4.0 mm lag screws, placed anteriorly to posteriorly. Fractures complicated by severe comminution necessitated 3.5 mm cortical screws in order to avoid shortening, translation or angulation of the fragments.
  Other Names: ORIF

SUMMARY:
The main purpose of this retrospective case series study was to evaluate long-term radiographic and clinical outcomes of a consecutive series of patients with diagnosis of isolated, displaced, closed talar neck or body fractures treated by open reduction and internal fixation. Secondly, it was aimed to verify the influence of the location of talar fractures on the outcomes, the prognostic value of the Hawkins sign, whether operative delays promote avascular necrosis (AVN) and if the fractures require emergent surgical management.

DETAILED DESCRIPTION:
From January 2007 to December 2012, 31 patients underwent ORIF by screws at our institution. On the basis of Inokuchi criteria, the injuries were divided between neck and body fractures, which were classified according to Hawkins and Sneppen, respectively. The patients included were divided into two groups in relation to fracture location and complexity. Radiographic assessment focused on reduction quality, bone healing, Hawkins sign and osteoarthritis development. For clinical evaluation, clinical-functional scores (AOFAS Ankle-Hindfoot Score; MFS; FFI-17; SF-36) and VAS were determined, and statistical analysis was performed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of a closed, isolated, displaced talar neck or body fracture with 2 or more millimetres displacement, subsequently treated by ORIF
* age between 18 and 85 years
* informed consent to participate.

Exclusion Criteria:

* undisplaced fractures or involvement of both the neck and the body,
* open fractures, talar head and peripheral fractures including posterior process, osteochondral fractures, primary arthrodesis or amputation,
* history of severe neurological deficit,
* previous foot surgery or trauma,
* diagnosis of rheumathological diseases or psoriatic arthritis, foot neuropathy, severe vascular insufficiency and alcohol or drug abuse.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There were 19 men (1 bilateral case for a total of 20 fractures, 71.4%) and 8 women (29.6%). Overall, mean age at the time of injury was 38.3 years old (range 18-81)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of the quality reduction after surgery | at day 1 after surgery
  Radiographic examination of anteroposterior, lateral and oblique view radiographs enabled to evaluate the quality of the reduction. Any offset of more than 2 mm or neck angulation of more than 5° between the fragment was labelled as a poor reduction.
Evaluation of bone healing | at different follow-ups (1 month, 3 months, 6 months, 12 months, 24 months)
  Criteria to define bone healing and union:
  The bridging bone/callus formation was evaluated on radiographs The absence of radiolucent lines was verified at different follow-ups.
Evaluation of osteonecrosis | at 6-8 weeks after injury
  The Hawkins sign appearance (only on the A/P X-ray), which resembles a subchondral atrophy in the talus dome, was evaluated indicating that the talus is well vascularized. On the contrary, its absence at this time suggests the presence of osteonecrosis
Evaluation of the development of post-injury peritalar osteoarthritis | at last follow-up (seven years)
  Post-injury peritalar osteoarthritis was evaluated on X-ray and differentiated between necrosis without collapse (sclerosis with and without geodes) and necrosis with collapse of the talar dome at the last follow-up

SECONDARY OUTCOMES:
American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot score | at last follow-up (seven years)
  The AOFAS score enabled to quantify pain and functional disability. It includes 9 questions related to pain (1 question; 40 points), function (7 questions; 50 points) and alignment (10 questions; 10 points); a score of 90-100 is considered an excellent result; 75-89 as good; 50-74 as fair and less than 49 points is considered a failure or a poor outcome.
the Maryland Foot Score (MFS) | at last follow-up (seven years)
  The MFS is a score conceptually analogous to AOFAS score, but points are differently distributed (45 for pain, 55 for functional limitation); they indicate excellent results if the score is between 90 to 100, good for a score of 75 to 89, fair for a score of 50 to 74 and poor if the score is < 50.
the 17-Foot Functional Index (FFI-17) | at last follow-up (seven years)
  The FFI-17 measures the persistence of pain, disability and restriction of activity, with 17 number-rating scales from 0 to 10. The maximum score is 100, which indicates complete disability.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Biz, MD, Principal Investigator — Padua University Orthopaedic Clinic

IPD SHARING:
Plan to Share IPD: No